CLINICAL TRIAL: NCT02195726
Title: The EUROpean and Asian Cardiac and Renal Remote Ischemic Pre-conditioning Study : A Prospective, Randomized Control Trial
Brief Title: Efficacy of RIPC to Reduce AKI for Patients Undergoing PCI
Acronym: EUROCRIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Claudio Moretti, Dottor, Head of the Catch Lab, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201301
Record Dates: First submitted 2013-01-14; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham remote ischemic preconditioning' (Sham Comparator): In the control group Sham remote ischemic preconditioning will be performed with inflation of 10 mmHg more than baseline
  Interventions: Procedure: Sham remote ischemic preconditioning
- Remote ischemic preconditioning (Experimental): In the experimental group, patients will receive for four times 5-minute inflations of a blood pressure cuff to 200 mmHg around the upper non dominant arm (or if systolic pressure is more than 150 mmHg, inflation will reach 50 mmHg upper than baseline), followed by 5-minute intervals of reperfusion.
  In subjects presenting with BMI > 30 a dedicated blood pressure cuff for obese patients will be used. Coronary angiography will be performed in 45 minutes from last inflation
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — four times 5-minute inflations of a blood pressure cuff to 200 mmHg around the upper non dominant arm (or if systolic pressure is more than 150 mmHg, inflation will reach 50 mmHg up per than baseline), followed by 5-minute intervals of reperfusion.
  Arms: Remote ischemic preconditioning
Procedure: Sham remote ischemic preconditioning — In the control group sham preconditioning will be performed with inflation of 10 mmHg more than baseline.
  Arms: Sham remote ischemic preconditioning'

SUMMARY:
The purpose of the present study is to determine if remote ischemic preconditioning reduces incidence of acute kidney injury in patients with reduced kidney function undergoing Percutaneous Coronary Intervention.

DETAILED DESCRIPTION:
Acute kidney injury negatively impacts on prognosis after PCI, and only hydratation have shown to reduce this complication.

Remote ischemic preconditioning has been demonstrated to reduce periprocedural MI, while impact on aki remains to be assessed

ELIGIBILITY:
Inclusion Criteria:

* undergoing PCI with stenting for all clinical indications
* carrying (with) a renal clearance less than 60 mL/min/1.73 m2 and more than 30 mL/min/1.73 m2 (evaluated through MDRD); ù
* younger than 85 years old.

Exclusion Criteria:

* ST Segment Elevation Myocardial Infarction (STEMI), unstable hemodynamic presentations (cardiogenic shock) or ongoing severe arrhythmias;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1110 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | 24 and 48 hours after PCI
  Acute Kidney Injury defined as Acute kidney injury is defined as an increase serum creatinine greater than 0.5 mg/dL, or by a relative increase of at least 25% over the baseline value within a period of 48-hours after contrast medium administration

SECONDARY OUTCOMES:
Incidence of periprocedural myocardial infarction | 24 and 48 hours after PCI

CONTACTS AND LOCATIONS:
Locations (7):
- Institut Cardiovasculaire Paris Sud Hôpital Jacques Cartier, Paris, France
- Italy (5):
  - Unità Operativa di Cardiologia Presidio Ospedaliero Misericordia Via Senese 161 58100 Grosseto, Grosseto
  - Azienda Ospedaliere Senese Siena, Siena
  - Ospedale Maria Vittoria, Turin
  - San Luigi, Turin
  - Città Della Salute e Della Scienza, Turin
- Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Derived] D'Ascenzo F, Femmino S, Ravera F, Angelini F, Caccioppo A, Franchin L, Grosso A, Comita S, Cavallari C, Penna C, De Ferrari GM, Camussi G, Pagliaro P, Brizzi MF. Extracellular vesicles from patients with Acute Coronary Syndrome impact on ischemia-reperfusion injury. Pharmacol Res. 2021 Aug;170:105715. doi: 10.1016/j.phrs.2021.105715. Epub 2021 Jun 7. PMID 34111564
- [Derived] Moretti C, Cerrato E, Cavallero E, Lin S, Rossi ML, Picchi A, Sanguineti F, Ugo F, Palazzuoli A, Bertaina M, Presbitero P, Shao-Liang C, Pozzi R, Giammaria M, Limbruno U, Lefevre T, Gasparetto V, Garbo R, Omede P, Sheiban I, Escaned J, Biondi-Zoccai G, Gaita F, Perl L, D'Ascenzo F. The EUROpean and Chinese cardiac and renal Remote Ischemic Preconditioning Study (EURO-CRIPS CardioGroup I): A randomized controlled trial. Int J Cardiol. 2018 Apr 15;257:1-6. doi: 10.1016/j.ijcard.2017.12.033. PMID 29506674
- See also: our research website group — http://www.cardiogroup.org/index.php?cat=home